#### Janssen Research & Development

#### **Statistical Analysis Plan**

A Randomized, Multicenter, Double-Blind, Parallel, Placebo-Controlled Study of the Effects of JNJ-28431754 on Cardiovascular Outcomes in Adult Subjects with Type 2 Diabetes Mellitus

The CANVAS Trial (CANagliflozin cardioVascular Assessment Study)

**Protocol 28431754DIA3008; Phase 3** 

JNJ-28431754 (canagliflozin)

**Status:** Approved

**Date:** 20 March 2017

**Prepared by:** Janssen Research & Development, LLC

**Document No.:** EDMS-ERI-130802595, 2.0

**Compliance:** The study described in this report was performed according to the principles of Good Clinical Practice (GCP).

#### **Confidentiality Statement**

The information in this document contains trade secrets and commercial information that are privileged or confidential and may not be disclosed unless such disclosure is required by applicable law or regulations. In any event, persons to whom the information is disclosed must be informed that the information is privileged or confidential and may not be further disclosed by them. These restrictions on disclosure will apply equally to all future information supplied to you that is indicated as privileged or confidential.

# **TABLE OF CONTENTS**

| TABLE | OF CONTENTS | . <b>2</b> |
|---|---|---|
| LIST O | F IN-TEXT TABLES | . 3 |
| LIST O | F IN-TEXT FIGURES | . 3 |
| SUMMA | ARY OF AMENDMENT | . 4 |
| ABBRE | VIATIONS | . 5 |
| 1. IN | TRODUCTION | . 6 |
| 1.1. | Trial Design | . 6 |
| 1.2. | Randomization | . 8 |
| 1.3. | Trial Objectives | . 8 |
| 1.3.1. | Primary Objectives | . 8 |
| 1.3.2. | Secondary Objectives | |
| 1.3.3. | Exploratory Objectives | |
| 1.4. | Statistical Hypotheses | 10 |
| 2. G | ENERAL ANALYSIS DEFINITIONS | 10 |
| 2.1. | Analysis Populations | 10 |
| | Analysis Sets | |
| 2.3. | Data Handling | |
| 2.3.1. | Censoring Rules | |
| 2.3.2. | Handling of Key Milestone Dates | |
| 2.3.3. | Visit Windows | |
| 3. SI | JBJECT INFORMATION | 40 |
| 3.1. | Baseline Anthropometric and Demographic Characteristics | |
| 3.1.<br>3.2. | Baseline Disease Characteristics | |
| 3.2.<br>3.3. | | |
| 3.4. | Disposition Information | |
| 3. <del>4</del> .<br>3.5. | Prior and Concomitant Medications | |
| 3.5. | Filor and Conconitant Medications | 15 |
| | FFICACY | |
| 4.1. | Primary Efficacy Endpoint | 16 |
| 4.1.1. | Definition | 16 |
| 4.1.2. | Analysis Methods | 16 |
| 4.1.3. | Subgroup Analyses | 17 |
| 4.1.4. | Supportive Analyses | |
| 4.1.4.1. | On-Study Analysis | |
| 4.1.4.2. | On-Treatment Analysis | |
| 4.1.4.3. | Additional Supportive Analyses | |
| 4.1.4.3. | , , | |
| 4.1.4.3. | | |
| 4.1.4.3. | | |
| 4.2. | Secondary Efficacy Endpoints | |
| 4.2.1. | Definition | |
| 4.2.2. | Analysis Methods | |
| 4.2.2.1. | | |
| 4.2.2.2. | Progression of Albuminuria | |
| 4.2.2.3. | Additional Secondary Endpoints | |
| 4.3. | Multiplicity Adjustment. | |
| 4.4. | Exploratory Efficacy Endpoints | 22 |
| 4.4.1. | Definition | |
| 4.4.2. | Analysis Methods | 23 |

| 4.4.2.1. | CV End | lpoints | 23 |
|---|---|---|---|
| 4.4.2.2. | | se Mortality | |
| 4.4.2.3. | | Endpoints | |
| 4.4.2.3.1. | | posite Endpoints | |
| 4.4.2.3.2. | | ression of Albuminuria | |
| 4.4.2.3.3. | | ession of Albuminuria | |
| 4.4.2.3.4. | | R Slope | |
| | • | | |
| | ETY | | <b>25</b> |
| 5.1. Ad | djudicated | I MACE Events | 25 |
| 5.2. Ad | dverse Ev | ents | 25 |
| 5.2.1. | Adverse E | Event Collection | 25 |
| 5.2.2. | Analysis I | Methods | 26 |
| 5.2.2.1. | Genera | I Adverse Events | 27 |
| 5.2.2.2. | Male M | ycotic Genital Infections | 28 |
| 5.2.2.3. | | ,<br>ycemia | |
| 5.2.2.4. | | d Malignancies | |
| 5.2.2.5. | | ensitivity | |
| 5.2.2.6. | Venous | Thromboembolic Events | 31 |
| 5.2.2.7. | | e | |
| 5.2.2.8. | | tion | |
| 5.2.2.9. | | C Ketoacidosis | |
| 5.2.2.10. | | atitis | |
| | | oratory Tests | |
| | | Oratory Tests | |
| | | iogram | |
| 0.0. Li | Collocala | logiani | 00 |
| REFEREN | ICES | | 36 |
| APPENDI | v | | 27 |
| | | List of Kou Anglings of OV and Martellity Endocints | |
| Appendix | | List of Key Analyses of CV and Mortality Endpoints | 3/ |
| Appendix | | Clinical Laboratory Tests | |
| Appendix | | Pre-defined Limit of Change (PDLC) Criteria | |
| Appendix | | List of Preferred Terms for Selected AEs of Interest | |
| Appendix | 1.5: | Adverse Events with Potential Amputation Association | 49 |
| LICTOF | · INI TEV | T TARLES | |
| LIST OF | IIN-I EX | T TABLES | |
| Table 1: | Summar | ry of Analysis Sets | 11 |
| Table 2: | Time Int | ervals for Analysis (in clinic) Visit Windows | 13 |
| Table 3: | Adverse | Events of Interest | 26 |
| Table 4: | | Factors Included in the Logistic Regression Analysis | |
| LIST OF | IN-TEX | T FIGURES | |
| | | | _ |
| Figure 1: | Diagram | of Study Designp of Randomized Subjects with Respect to the GTED | / |
| i iquit 2. | i UllUW-U | ID OF NATIOUTIES OUD SOLD WITH INCODES TO THE OFFI | 0 |

# **SUMMARY OF AMENDMENT**

Relative to the statistical analysis plan (SAP) dated 20 September 2016, the major amendments made in this version are summarized as follows.

| Applicable | |
|---|---|
| Section(s) | Description of Change(s) |
| 1.3.3 | Removed 'Change in eGFR from baseline to the last off-drug value' from |
| 4.4 | objectives and exploratory efficacy endpoints. |
| 2.2 | The On-Study analysis set was added for MACE and replaced the ITT analysis set for several adverse events of interest. The upper bound of the data period for the On-Treatment analysis set was clarified as last dose plus 2 days for laboratory parameters except ACR. |
| 4.1 | Consistent with the analytic approach described in the Cardiovascular Endpoint adjudication charter, it is clarified that undetermined death is considered as CV death. |
| 4.1.3 | Additional subgroups were added for the analysis of MACE. |
| 4.1.4.3.1 | Added an analysis of MACE in the first 30, 60 and 90 days. |
| 4.1.4.3.3 | Updated the multiple imputation analysis section |
| 4.2 | Added analysis based on MMRM for continuous secondary efficacy endpoints. |
| 4.4 | Clarified that any adjudicated non-CV death event where the adjudication committee assigned a renal proximate cause is considered a renal death. |
| 5.2.2.10 | Added a section on the analysis of adjudicated pancreatitis. |
| Appendix 1.3 | Additional lab analytes were included in the Pre-defined Limit of Change (PDLC) criteria. |

#### **ABBREVIATIONS**

ACR albumin creatinine ratio

AE adverse event

AHA antihyperglycemic agent ANCOVA analysis of covariance

BL baseline

BMI body mass index

CHMP Committee for Medicinal Products for Human Use

CI confidence interval CV cardiovascular

DBP diastolic blood pressure DKA diabetic ketoacidosis

EAC Endpoint Adjudication Committee

eCRF electronic case report form

eGFR estimated glomerular filtration rate FDA Food and Drug Administration

FPG fasting plasma glucose GTED Global Trial End Date  $HbA_{1c}$  hemoglobin  $A_{1c}$ 

HDL-C high-density lipoprotein cholesterol

HR hazard ratio

IDMC independent data monitoring committee

ITT intent-to-treat

IWRS interactive web response system LDL-C low-density lipoprotein cholesterol

LLN lower limit of normal

MACE major adverse cardiovascular event

MedDRA Medical Dictionary for Regulatory Activities

MI myocardial infarction
PDLC pre-defined limit of change

PT preferred term

QTcF QTc using the Fridericia

RAAS renin angiotensin aldosterone system

SAE serious adverse event
SAP statistical analysis plan
SBP systolic blood pressure
SC steering committee
SCr serum creatinine
SD standard deviation

SGLT2 sodium-glucose co-transporter 2

SI standard international
SOC System Organ Class
T2DM type 2 diabetes mellitus
TEAE treatment-emergent AE
ULN upper limit of normal
UTI urinary tract infection

VTE venous thromboembolic events

#### 1. INTRODUCTION

Canagliflozin (JNJ-28431754) is an inhibitor of the sodium-glucose co-transporter 2 (SGLT2) that has been developed as an oral anti-hyperglycemic agent (AHA) for the treatment of patients with type 2 diabetes mellitus (T2DM). To meet the FDA guidance on assessing cardiovascular (CV) safety of AHAs, the sponsor initiated the CV outcomes study 28431754DIA3008 (CANVAS) in December, 2009 intended to supply data to support the CV safety of canagliflozin and to also evaluate whether canagliflozin reduces CV risk.

As part of the marketing authorization application, the sponsor performed an integrated analysis of CV events from the Phase 2 and Phase 3 canagliflozin program using data from 9,632 subjects, which included interim data harvested on 31 January 2012 from the ongoing CANVAS study of 4,330 subjects at high risk for CV disease. Subsequently, in response to a request arising during review of the canagliflozin Marketing Authorization Application by the Committee for Medicinal Products for Human Use (CHMP), the sponsor conducted a second integrated CV analysis of the Phase 2 and Phase 3 studies, which included interim data from CANVAS harvested on 19 November 2012. Data on major adverse cardiovascular events (MACE) and mortality outcomes beyond 19 November 2012 have remained blinded to the sponsor.

The primary endpoint of CANVAS was to evaluate whether there was a risk reduction in MACE associated with canagliflozin treatment. Due to unblinding of the interim summary results of CANVAS at the time of marketing approval, the planned expansion of enrollment in CANVAS was eliminated. Accordingly, the study itself is underpowered for the primary hypothesis of the reduction in CV risk as measured by the hazard ratio (HR) for MACE.

As a result of the discussions with FDA, the sponsor proposed to conduct a second CANVAS-like study (referenced as CANVAS-R) with approximately 5,700 randomized subjects. As such, the CANVAS and CANVAS-R trials are purposefully similar in design and in subject characteristics. Data from these studies are to be harvested for an integrated analysis to meet the FDA post-approval CV safety requirement and if safety is demonstrated, to assess whether canagliflozin reduces all-cause mortality no later than June 2017 with study reports submitted to FDA by September 2017.

This statistical analysis plan (SAP) stipulates definitions of analysis sets, key derived variables and statistical methods for analysis of efficacy and safety specific for CANVAS based on the latest amendment INT-8 (5 May 2016) of the protocol. Additional CV and renal outcome endpoints are added in this SAP for exploratory analysis. Since the Clinical Study Reports of the 18-week substudies were submitted in the NDA of canagliflozin and the 52-week interim results were published, the analyses in these sub studies will not be addressed in this plan.

#### 1.1. Trial Design

The CANVAS study enrolled the first subject in December 2009. The original design called for the study to be conducted in 2 cohorts (an initial cohort of 4,500 subjects enrolled prior to regulatory submissions followed by a subsequent cohort of 14,000 subjects to be enrolled post approval).

However, due to unblinding of the interim summary results of CANVAS at the time of marketing approval, the planned expansion of enrollment in CANVAS was eliminated.

The study enrolled 4,330 subjects who met all inclusion criteria and none of the exclusion criteria. Subjects were randomly assigned to treatment with 1 of 2 doses of canagliflozin (100 or 300 mg) or placebo, in a 1:1:1 ratio. The CANVAS and CANVAS-R studies will complete when the last subject randomized has approximately 78 weeks of follow-up or when 688 MACE events are accumulated between both studies (estimated to occur between January 2017 and April 2017). The announcement of the Global Trial End Date (GTED) will mark the anticipated date on which one of these requirements for ending the study will occur.

Following announcement of the projected GTED and for subjects remaining on double-blind study drug, sites will schedule the End of Treatment (EOT) and the 30-day off-drug follow-up contact as per the Time and Events schedule in the protocol; for subjects that have prematurely discontinued study drug prior to the announcement of the projected GTED, sites will be required to make a final contact or vital status check as soon as possible after the announcement of the GTED.

A single Steering Committee (SC) and an Independent Data Monitoring Committee (IDMC) are commissioned for this and the CANVAS-R study. The SC oversees the study conduct, and the IDMC regularly (and on an ad hoc basis) reviews safety data.

Figure 1 shows an overview of the study design and Figure 2 shows the scheduled follow-up of randomized subjects prior to the GTED.



AHA=antihyperglycemic agent; CV=cardiovascular; HbA<sub>1c</sub>=hemoglobin A<sub>1c</sub>; GTED=global trial end date; R=randomization; SU=sulfonylurea; T2DM=type 2 diabetes mellitus



Figure 2: Follow-up of Randomized Subjects with Respect to the GTED

Note: Following the announcement of the GTED, investigators are not expected to continue collecting data for purposes of the clinical trial after the 30-day post-treatment contact.

#### 1.2. Randomization

Subjects were stratified into one of 6 predefined strata based on AHA use at the run-in visit through to the randomization visit. The investigators were instructed to hold AHA use constant through Week 18 and to adjust the subject's AHA regimen after Week 18 so as to achieve target glycemic control throughout the remainder of the study.

Central randomization was implemented in this study. Subjects were randomly assigned to 1 of 3 treatment groups based on a computer-generated randomization schedule prepared by the sponsor before the study. The randomization was balanced by using randomly permuted blocks and was stratified based on the use of specific concomitant AHA medications at baseline.

# 1.3. Trial Objectives

#### 1.3.1. Primary Objectives

In subjects with T2DM, with inadequate glycemic control, who have a history or high risk of CV disease:

- To assess the effect of canagliflozin plus standard of care relative to placebo plus standard of care on CV risk as measured by the HR for a composite endpoint (MACE including CV death, nonfatal MI, or nonfatal stroke);
- To assess the safety and tolerability of canagliflozin plus standard of care relative to placebo plus standard of care.

# 1.3.2. Secondary Objectives

In subjects with T2DM, with inadequate glycemic control, who have a history or high risk of CV disease, to assess the effect of canagliflozin plus standard of care relative to placebo plus standard of care at the end of the treatment period on:

- Fasting measures of beta-cell function (HOMA-B and the proinsulin/insulin ratio) (note: this assessment will be conducted in a subset of subjects at sites that elected to participate, including only subjects who did not receive insulin at randomization);
- The proportion of subjects with progression of albuminuria (progression defined as the development of microalbuminuria or macroalbuminuria in a subject with baseline microalbuminuria);
- Urinary albumin/creatinine ratio (ACR);
- Change from baseline in estimated glomerular filtration rate (eGFR);
- Change from baseline in HbA<sub>1c</sub> and fasting plasma glucose (FPG);
- Change in body weight;
- Change in blood pressure (systolic and diastolic);
- Change in fasting plasma lipids (triglycerides, high-density lipoprotein cholesterol [HDL-C], low-density lipoprotein cholesterol [LDL-C], total cholesterol, and the ratio of LDL-C to HDL-C).

# 1.3.3. Exploratory Objectives

In subjects with T2DM, with inadequate glycemic control, who have a history or high risk of CV disease, to assess the effect of canagliflozin plus standard of care relative to placebo plus standard of care on:

- Hospitalization for heart failure;
- The composite of hospitalization for heart failure or CV death;
- The composite of 40% decrease in eGFR, renal death or requirement for renal replacement therapy;
- The composite of doubling of serum creatinine (SCr), renal death or requirement for renal replacement therapy;
- The composite of 40% decrease in eGFR, renal death, requirement for renal replacement therapy or CV death;
- The composite of doubling of SCr, renal death, requirement for renal replacement therapy or CV death;
- The composite of 40% decrease in eGFR, conversion to macroalbuminuria, renal death or requirement for renal replacement therapy;
- The composite of doubling of SCr, conversion to macroalbuminuria, renal death or requirement for renal replacement therapy;

- Progression of albuminuria (defined as the development of microalbuminuria or macroalbuminuria in a subject with baseline normoalbuminuria or the development of macroalbuminuria in a subject with baseline microalbuminuria), accompanied by an ACR value increase of greater than or equal to 30% from baseline;
- Regression of albuminuria (regression defined as the development of normoalbuminuria in a subject with baseline microalbuminuria or macroalbuminuria or the development of microalbuminuria in a subject with baseline macroalbuminuria), accompanied by an ACR value decrease of greater than or equal to 30% from baseline;
- Change in eGFR determined from a between-group comparison of the eGFR slopes using all on-drug measurements (ie, off-drug values will not be included) of eGFR made from the first on-drug measurement to the final on-drug measurement.

# 1.4. Statistical Hypotheses

The following hypotheses are specified in the study protocol, however they are considered to be exploratory in the canagliflozin CV outcome consisting of CANVAS and CANVAS-R. The hypotheses in this trial are not included as part of the testing sequence of the program. Accordingly, any p-value reported will be considered as nominal and 95% confidence intervals (CIs) for the treatment effect will be presented for descriptive purposes.

In subjects with T2DM with inadequate glycemic control, who have a history of or a high risk of CV disease, relative to placebo plus standard of care, canagliflozin plus standard of care:

- Reduces CV risk (as measured by the HR for MACE including CV death, nonfatal MI, and nonfatal stroke);
- Improves beta-cell function (change from baseline in HOMA-B) at the end of the treatment period;
- Reduces progression of albuminuria (ie, proportion of subjects with a  $\geq 1$ -step progression of albuminuria measured by the urine ACR) at the end of the treatment period.

#### 2. GENERAL ANALYSIS DEFINITIONS

# 2.1. Analysis Populations

- Randomized subjects—subjects who are randomized via the Interactive Web Response System (IWRS);
- Treated subjects—randomized subjects who received at least one dose of double-blind study medication.

For efficacy analyses and baseline summaries, subjects will be analyzed according to their randomization assignment. For safety analyses (eg, adverse events [AEs]) and the summary of exposure, subjects will be analyzed according to the predominant treatment received (defined as the treatment to which the subject was exposed for the greatest duration), in the event that subjects receive a treatment other than the one to which they were randomized.

# 2.2. Analysis Sets

Analysis sets consist of 2 components: 1) analysis population (Section 2.1), which specifies the subjects included in an analysis; 2) data period, defining the time window during which data will be included in the analysis.

Safety data collection in CANVAS was streamlined after protocol amendment INT-6 (effective starting on 07 January 2014) such that AEs were only collected if they were serious or leading to study drug discontinuation, with the exception of selected AEs of interest. For the purpose of summarizing safety data *prior* to amendment INT-6, the On-Treatment Pre-INT6 analysis set was created as described below.

**Table 1:** Summary of Analysis Sets

| Analysis Set | Analysis Population | Data Period |
|---|---|---|
| ITT | Randomized subjects | |
| 1111 | Randomized subjects | Day 1 to the last trial contact date (refer to |
| | | Section 2.3.2) up to the GTED |
| On-Study | Treated subjects | Day 1 to the last trial contact date (see Section 2.3.1) |
| _ | | up to GTED |
| On-Treatment | Treated subjects | Day 1 to the last dose date (refer to Section 2.3.2) plus |
| | | X <sup>a</sup> days or the last trial contact date, whichever is |
| | | earlier |
| On-Treatment | Treated subjects | Day 1 to the last dose date plus X <sup>a</sup> days or the last trial |
| Pre-INT6 | | contact date, whichever is earlier, up to |
| | | 07 January 2014 |

X is 2 days for laboratory (except ACR) and vital sign measurements, and 30 days for CV and mortality endpoints, and adverse events.

# 2.3. Data Handling

#### 2.3.1. Censoring Rules

For each analysis set, events that occur any time during the data period of the corresponding analysis set (refer to Table 1) will be considered as eligible events; otherwise subjects not experiencing an event will be censored at the earlier of the last trial contact date or end of the respective data period, if not otherwise specified.

#### 2.3.2. Handling of Key Milestone Dates

- Trial reference start date (Day 1): the first double-blind dose date for each subject (First dose date). If missing or incomplete, the first dose date will be imputed as the randomization date.
- Last dose date: the date on which the last dose of double-blind study drug was taken by the subject. If only the day is missing, impute the last day of the month. If the month or the year is missing, impute the date as the date of the scheduled visit subsequent to the last visit when the study drug was dispensed. The imputed last dose date should be no later than the end of treatment visit date or the last trial contact date. In addition, the imputed last dose date should be no earlier than the first dose date. The last dose date is the date of permanent study drug discontinuation regardless of any temporary drug interruption.

- Last trial contact date: the date when the last trial-related procedure is conducted. It is defined as the latest of:
  - The date of last visit (scheduled or unscheduled visit; office or phone visit), or
  - The latest known date of an AE or the study endpoint event status, concomitant medication, vital sign measurements or laboratory results as reported on their respective electronic case report form (eCRF), or
  - The date of alternate contact made (eg, family members, relatives, friends, health care providers, public search) confirming the subject's survival status at the time of the GTED.
  - For subjects who die during the study, the last trial contact date will be defined as the date of death.

### 2.3.3. Visit Windows

The Time and Events schedule of the protocol indicates the visit timing and procedures (eg, laboratory, vital signs, and other key safety variables) for each visit; however, the timing of a subject's actual visit may not be exactly as per the protocol indicated target day / visit window. Consequently, for by-visit or over-time summaries, depending on the time period(s) involved in the summaries, the conventions outlined below will be used to allocate the data collected at each actual visit to a planned protocol visit by defining visit windows.

Baseline will be defined as the pre-dose measurement closest to or including Day 1 (prior to dose administration). If the pre-dose measurement on Day 1 is missing, the missing value will be imputed by the latest available measurement prior to Day 1.

If a subject has 2 or more actual visits in one analysis visit window, the visit closest to the target day will be used as the study visit for that analysis visit window. However, results from all visits will be included in the safety analyses (eg, pre-defined limits of change analysis) to assure that all results are included. If 2 study visits are the same number of days from the target day within the same visit window, the later visit will be considered the study visit for that target day. Even though all visits will be allocated an analysis visit window, only planned protocol visits for each variable will be included in the by-visit summaries or repeated measure analyses.

Note that the algorithms for calculating visit windows are the same for all the data periods (refer to Table 1). Table 2 summarizes the analysis visit windows for laboratory, vital signs, and other key safety variables.

| Table 2: | Time Intervals for . | Analysis (in clinic | Visit Windows |
|----------|----------------------|---------------------|---------------|
|----------|----------------------|---------------------|---------------|

| Scheduled Visit Time | Time Interval | Target Time |
|----------------------|--------------------|-------------|
| (label on output) | (Day) <sup>a</sup> | Point (Day) |
| Baseline | ≤1 <sup>b</sup> | 1 |
| Week 6 | 1°-64 | 43 |
| Week 12 | 65 – 99 | 85 |
| Week 18 | 100 – 155 | 127 |
| Week 26 | 156 – 197 | 183 |
| Week 39 | 198 – 288 | 274 |
| Week 52 | 289 – 456 | 365 |
| Week 78 | 457–638 | 547 |
| Week 104 | 639–820 | 729 |
| Week 130 | 821–1002 | 911 |
| Week 156 | 1003-1184 | 1093 |
| Week 182 | 1185–1366 | 1275 |
| Week 208 | 1367–1548 | 1457 |
| Week 234 | 1549 – 1730 | 1639 |
| Week 260 | 1731 – 1912 | 1821 |
| Week 286 | 1913 – 2094 | 2003 |
| Week 312 | 2095 – 2276 | 2185 |
| Week 338 | 2277 – 2458 | 2367 |
| Week 364 | 2459 – 2640 | 2549 |
| Week 390 | 2641 – 2822 | 2731 |

<sup>&</sup>lt;sup>a</sup> Relative to the day of the first dose of double-blind study drug.

#### 3. SUBJECT INFORMATION

# 3.1. Baseline Anthropometric and Demographic Characteristics

Baseline anthropometric and demographic characteristics will be summarized by treatment group (each canagliflozin dose and all canagliflozin group, as well as placebo). Descriptive statistics (N, mean, standard deviation, median, and range) will be provided by treatment group for baseline age and baseline body weight.

Additionally, the number and percentage of subjects in the categories of the following variables at baseline will also be summarized by treatment group:

- Age group:  $<65, \ge 65$  years old;
- Sex: Male, Female;
- Race: White, Black or African American, Asian, Others;
- Ethnicity: Hispanic or Latino, Not Hispanic or Latino, Unknown, Not reported;
- Region: North America, Central/South America, Europe, Rest of the World.

b Up to the first dose of double-blind study drug.

Immediately following the first dose of double-blind study drug. For variables with no time or reference collected at baseline, the first window after baseline starts on Day 2 according to the protocol.

#### 3.2. Baseline Disease Characteristics

Descriptive statistics (N, mean, SD, median, and range) will be provided by treatment group and overall for the following baseline continuous variables: duration of diabetes (in years), eGFR, ACR, systolic blood pressure (SBP), weight, body mass index (BMI), HbA<sub>1c</sub>, LDL-C, HDL-C, triglycerides, total cholesterol, and LDL-C/HDL-C.

Additionally, the number and percentage of subjects will be summarized by treatment group and overall for the following:

- Baseline BMI categories (<30, ≥30 kg/m²);
- Currently daily cigarette smoker: Yes/No;
- Baseline  $HbA_{1c} \ge 8\%$ : Yes/No;
- Duration of T2DM  $\geq$  10 years: Yes/No;
- Baseline systolic blood pressure categories (≤140, >140 mmHg);
- Baseline LDL-C categories ( $\leq 70$ , > 70 mg/dL);
- Baseline HDL-C categories (<39,  $\ge39$  mg/dL);
- Baseline eGFR categories (<30, 30 to <60, 60 to <90, ≥90 mL/min/1.73m<sup>2</sup>);
- Baseline albuminuria categories:
  - Normoalbuminuria (0 ≤ ACR <30 mg/g); Microalbuminuria (ACR ≥30 mg/g and  $\leq$ 300 mg/g); Macroalbuminuria (ACR > 300 mg/g: ACR >300 mg/g and  $\leq$ 3000 mg/g, ACR > 3000 mg/g).
- History of hypertension: Yes/No;
- History of CV disease: Yes/No;
- History of coronary artery disease: Yes/No;
- History of cerebrovascular disease: Yes/No;
- History of peripheral vascular disease: Yes/No;
- History of heart failure: Yes/No;
- Microvascular diabetes complications (Any, 1, 2 or 3 of retinopathy, neuropathy [diabetic or autonomic neuropathy] and nephropathy);
- History of fracture: Yes/No;

The number and percentage of subjects with a history of medical conditions by system organ class and preferred term (based upon the general medical history eCRF) will be summarized by treatment group and overall.

# 3.3. Disposition Information

Disposition will be summarized for all randomized subjects by treatment group using the categories listed below:

- Screen failure;
- Subjects who are randomized (ITT);
- Subjects who are treated;
- Subjects who complete the study (ie, defined as having been followed until a time point between the notification of the GTED and the GTED, or if the subject has died prior to the GTED);
- Subjects who prematurely discontinued study medication;
- Subjects without final vital status.

The reasons for non-randomization, withdrawal from study (eg, lost to follow-up, consent withdrawal), and discontinuation from study medication will be summarized. The distribution of time to premature discontinuation of study medication will be displayed using a Kaplan-Meier plot, where one minus the survival function will be shown.

Listings will be provided for subjects whose predominant treatment differs from their randomized treatment.

# 3.4. Extent of Exposure and Follow-Up

Total exposure time for each subject is defined as the number of days from Day 1 to the last dose date (inclusive), regardless of any temporary drug interruption(s). Follow-up time is defined as the number of days from Day 1 to the last contact day (inclusive) for each subject. Descriptive statistics (N, mean, SD, median, and range) for total exposure or follow-up time will be presented by treatment group.

The number of subjects with duration in each of the following categories (<3 week, 3 to <13 week, 13 to <26 weeks, 26 to <52 weeks, 52 to <78 weeks, 78 to <104 weeks, 104 to <130 weeks, 130 to <156 weeks, 156 to <182 weeks, 182 to <208 weeks, 208 to <234 weeks, 234 to <260 weeks, 260 to <286 weeks, 286 to <312 weeks, 312 to <338 weeks, and  $\ge338$  weeks) will also be presented by treatment group as well as overall.

#### 3.5. Prior and Concomitant Medications

Concomitant medication usage is collected on the eCRF at baseline, and during the on-drug period. The number of subjects receiving medication in pre-specified categories will be presented by treatment group at baseline and on-drug period. In addition, SGLT2 inhibitor use during the off-drug follow-up period will also be summarized by treatment group.

All study medications are coded using World Health Organization Drug Utilization Research Group (WHODRUG) and Anatomical Therapeutic Chemical (ATC) codes.

Additionally, the number and percentage of subjects taking the following concomitant medications at baseline will be summarized by treatment group and overall:

- Baseline insulin use: Yes/No;
- Baseline sulphonylurea use: Yes/No;
- Baseline metformin use: Yes/No;
- Baseline statin use: Yes/No;
- Baseline anti-thrombotic use: Yes/No;
- Baseline diuretic use: Yes/No:
  - Baseline loop diuretic use: Yes/No;
  - Baseline non-loop diuretic use: Yes/No;
- Baseline renin angiotensin aldosterone system (RAAS) inhibitor use: Yes/No.

#### 4. EFFICACY

The primary analysis will be performed based on the ITT analysis set and secondary efficacy endpoints will be based on the On-treatment analysis set, if not otherwise specified.

As noted in Section 1, there will be no formal statistical hypothesis testing and therefore all statistical tests will be considered nominal and reported using a 2-sided 95% confidence level.

Unless otherwise stated, all efficacy analyses and summaries will be performed using the treatment groups assigned by IWRS.

A tabulation of all the key analyses planned for the CV endpoints and the mortality endpoint is presented in Appendix 1.1.

# 4.1. Primary Efficacy Endpoint

#### 4.1.1. Definition

The primary efficacy endpoint is the time to MACE (ie, composite of CV death<sup>a</sup>, non-fatal MI<sup>b</sup>, and non-fatal stroke), which is calculated as the time from Day 1 to the first occurrence of MACE. Adjudication of these outcomes by the Endpoint Adjudication Committee (EAC) will be done in a blinded fashion.

# 4.1.2. Analysis Methods

The primary analysis will be based on the ITT analysis set for adjudicated MACE. The HR of canagliflozin (all canagliflozin group as well as each canagliflozin dose) compared to placebo and

\_

<sup>&</sup>lt;sup>a</sup> Undetermined death is considered CV death.

<sup>&</sup>lt;sup>b</sup> Silent MIs are excluded from the analysis.

its 95% CI will be estimated using a stratified Cox proportional hazards model with a term for treatment as the explanatory variable and history of CV disease (secondary and primary prevention) as a stratification factor.

The percentage of subjects who experience a MACE and the corresponding incidence rate per 1,000 patient-years will be reported. The cumulative event rate over time will be presented using a Kaplan-Meier plot by treatment (all canagliflozin group and placebo as well as each canagliflozin dose and placebo).

#### 4.1.3. Subgroup Analyses

The homogeneity of treatment effect on the occurrence of the primary endpoint across subgroups will be examined (at a 2-sided significance level of 0.05) via a test for the treatment by subgroup interaction by adding this term and the subgroup as covariates (treated as class variables) to the primary efficacy analysis (Section 4.1.2) model. Subgroup analysis will be conducted when the total number of events is greater than 10 for two treatment groups (all canagliflozin group and placebo) and at least 1 event in both groups. Factors exhibiting interactions at a significance level of  $p \le 0.05$  will be identified as suggesting treatment effect heterogeneity, recognizing the multiplicity in testing multiple subgroups such that one or more p-values  $\le 0.05$  may be expected to be observed by chance alone.

If a significant interaction is observed, the Gail-Simon test will be used to further examine the nature of the interaction (qualitative or quantitative).

The HR of canagliflozin (all canagliflozin group) compared to placebo and its 95% CI will be estimated for each of the following subgroups:

- Age group:  $<65, \ge 65$  years old;
- Sex: Male, Female;
- Race: White, Black or African American, Asian, Other;
- Region: Central/South America, Europe, North America, Rest of the World;
- Baseline BMI categories (<30, ≥30 kg/m²);</li>
- Baseline composite blood pressure categories ([SBP<140or DBP<90 mmHg] vs. [SBP ≥140 and DBP ≥90 mmHg]);</li>
- Baseline eGFR categories (30 to <60, 60 to <90, ≥90 mL/min/1.73m<sup>2</sup>);
- Baseline  $HbA_{1c} \ge 8\%$ : Yes/No;
- Duration of diabetes ≥ 10 years: Yes/No;
- History of CV disease: Yes/No;
- History of peripheral vascular disease: Yes/No;
- History of amputation: Yes/No;
- Baseline use of statin;

- Baseline use of anti-thrombotics;
- Baseline use of RAAS inhibitor;
- Baseline use of Beta blocker;
- Baseline use of insulin;
- Baseline use of diuretics.

# 4.1.4. Supportive Analyses

If not otherwise specified, the supportive analyses will use the same analysis set as in the primary efficacy analysis.

# 4.1.4.1. On-Study Analysis

The stratified Cox proportional hazards model (as described in Section 4.1.2) will be repeated using the On-Study analysis set, in which data of treated subjects from Day 1 to the last trial contact date up to the GTED are used.

The percentage of treated subjects who experience a MACE and the corresponding incidence rate per 1,000 patient-years will be reported.

# 4.1.4.2. On-Treatment Analysis

The primary analysis (as described in Section 4.1.2) will be repeated using the On-Treatment analysis set, in which data from Day 1 to 30 days after the last dose of the study drug are used.

#### 4.1.4.3. Additional Supportive Analyses

#### 4.1.4.3.1. MACE in the First 30, 60 and 90 Days

In addition to the Kaplan-Meier plot described in Section 4.1.2, frequency counts (n and %) of subjects experiencing the first occurrence of MACE within the first 30 days, 60 days and 90 days will be provided in the ITT analysis set.

# 4.1.4.3.2. Hazard Ratio Estimation for Individual MACE Components

A separate analysis will be performed for each individual MACE component (CV death, nonfatal MI, or nonfatal stroke) in both the ITT analysis set and the On-Treatment analysis set. Additionally, analyses of fatal/non-fatal MI as well as fatal/non-fatal stroke will be performed. For subjects who experience more than one MACE component, all events will be counted in the analysis for the relevant component (eg, if a subject has both non-fatal MI and non-fatal stroke, the subject will be counted as having each event). The percentage of subjects who experience each MACE component and the corresponding incidence rate per 1,000 patient-years will be summarized by treatment. The HR of canagliflozin (all canagliflozin group as well as each canagliflozin dose) compared to placebo and its 95% CI will be estimated using a stratified Cox proportional hazards model with a term for treatment as the explanatory variable and history of CV disease (secondary and primary prevention) as a stratification factor.

# 4.1.4.3.3. Assessment of Missing Data

The impact of missing data in the interpretation of the primary efficacy analysis will be explored. For subjects who are lost to follow-up or withdrew consent before the development of a MACE in the ITT analysis set, data collected between the last trial contact date and the GTED will be considered missing.

The proportion of data missing, defined as the ratio of the duration of missing follow-up (eg, days between last contact date + 1 day and the GTED) and the duration of intended follow-up (eg, days between randomization date and the GTED) will be summarized.

#### **Multiple Imputation**

The estimate of interest is the hazard ratio to develop MACE among all randomized subjects regardless of adherence to study medication over the period between randomization and the global trial end date (GTED). For subjects who are lost to follow up or withdrew consent before the development of a MACE, data between the last trial contact date and the GTED will be considered missing.

The subjects who discontinued from study medication prematurely prior to the announcement of the GTED can have a different hazard from those who stay on treatment throughout the trial, and their corresponding drop-out could be considered informative. This subpopulation is defined to be the subjects who

- discontinued from study medication prior to the announcement of the GTED, and
- for whom death is not the reason for the discontinuation of study medication.

The data used to model imputed outcomes for subjects with missing data will be those of the subpopulation including the retrieved drop-out data. The definition of the retrieved drop-out data is the follow up data between treatment discontinuation and the GTED. Subjects who developed MACE prior to the treatment discontinuation are included in the subpopulation and their time to MACE data will be used for the imputation modeling. With these subjects included, the model estimate of hazard should fully reflect the potential hazard of the subjects with missing outcome.

A Weibull parametric time to event model (the imputation model) will be fit using the observed time to MACE data from the subpopulation described above. The model will be stratified by study and prior cardiovascular disease (Yes/No), and adjust for treatment and the following covariates potentially correlated with missing mechanism and risk of MACE so that bias due to informative censoring in the estimation of hazard could be minimized and the precision could be optimized.

- Completion of follow up to GTED: Yes/No
- Age group:  $<65, \ge 65$  years old;
- Sex: Male, Female;
- Baseline use of Metformin: Yes/No;

- History of heart failure: Yes/No;
- Baseline SBP >140 mmHg: Yes/No;
- Baseline  $HbA_{1c} \ge 8\%$ : Yes/No;

In case the model does not converge, covariates will be removed from the model in the descending order as listed.

For subjects with missing data, follow up time post drop-out will be imputed with random values derived from the conditional distribution of the missing data, given the observed data and the parameters estimated from the imputation model with the pre-specified covariates. If the sum of the observed time and the simulated time is less than the expected follow-up time, ie, from randomization to the GTED, an event is imputed for the corresponding subject. Otherwise, the subjects will be censored at GTED.

The imputed events and follow-up times will be integrated with the observed data. The primary efficacy model will be reanalyzed with the imputed dataset. This process will be repeated 1,000 times. The multiple analysis results will be combined into a single inferential summary (ie, HR and 95% CI) using Rubin's rules.<sup>1</sup>

#### 4.2. Secondary Efficacy Endpoints

#### 4.2.1. Definition

The secondary efficacy endpoints are:

- Change from baseline to the end of treatment in HOMA-B:
- The proportion of subjects with progression of albuminuria at the end of treatment (ie, the development of microalbuminuria or macroalbuminuria in a subject with baseline microalbuminuria);
- Change in proinsulin/insulin ratio:
- Change in urinary ACR;
- Change in eGFR;
- Change in HbA<sub>1c</sub>;
- Change in FPG;
- Percent change in body weight;
- Change in blood pressure (systolic and diastolic);
- Percent change in fasting plasma lipids (triglycerides, HDL-C, LDL-C, total cholesterol, and the ratio of LDL-C to HDL-C).

# 4.2.2. Analysis Methods

Unless otherwise specified, the analyses for the secondary efficacy endpoints will be using the On-Treatment analysis set. Only subjects with a baseline and at least 1 post-baseline measurement will be included in the analysis.

#### 4.2.2.1. HOMA-B

The analyses for beta-cell function will be conducted in a subset of subjects at sites that elected to participate, including only subjects who are not receiving insulin at randomization. For subjects who initiated insulin during the study, all HOMA-B data after the initiation of insulin will be censored.

Changes in HOMA-B from baseline will be analyzed using an analysis of covariance (ANCOVA) model with treatment as the explanatory variable and baseline HOMA-B value as a covariate. The treatment difference in the least-squares means and the 2-sided 95% CI will be estimated based on this model.

Change from baseline in HOMA-B over time will be analyzed using a mixed model for repeated measures (MMRM) based on restricted maximum likelihood (REML). The analysis will be based on observed data and will include the fixed, categorical effects of treatment, visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline and baseline-by-visit interaction. An unstructured covariance will be used to model the within-patient errors. The treatment comparison will be based on the least squares means and the 2-sided 95% CI will be estimated.

Descriptive statistics will be calculated for the change from baseline over time based on observed data.

#### 4.2.2.2. Progression of Albuminuria

The proportion of subjects with progression of albuminuria at the end of treatment will be analyzed using the logistic model with treatment as the explanatory variable and baseline albuminuria status as a covariate. Subjects without baseline and/or post-baseline ACR measurements will be excluded from the analysis. Furthermore, subjects with macroalbuminuria at baseline (ACR >300 mg/g) will also be excluded from the analysis. Baseline ACR value is derived as the geometric mean of all predose ACR measurements. For ACR values below the lower quantifiable limit, the lower quantifiable limit itself will be used for analysis. The odds ratios and the 2-sided 95% CIs for the treatment comparisons will be derived from the model. Albuminuria will be assessed according to the categorizations defined in the National Kidney Foundation Kidney Disease Outcomes Quality Initiative Guideline #1:<sup>2</sup> microalbuminuria is defined as ACR of 30 to 300 mg/g and macroalbuminuria is defined as an ACR greater than 300 mg/g.

Data obtained up to last dose plus 30 days will be included this analysis.

# 4.2.2.3. Additional Secondary Endpoints

The analyses for the additional secondary efficacy endpoints will be based on the On-Treatment analysis set. Only subjects with baseline and at least one post-baseline measurement will be included in the analysis.

Changes at the end of treatment from baseline in proinsulin/insulin ratio, eGFR, HbA<sub>1c</sub>, FPG, blood pressure, percent change in body weight and fasting lipids (HDL-C, LDL-C, triglycerides, total cholesterol, and LDL-C/HDL-C) will be analyzed using an analysis of covariance (ANCOVA) model with treatment and the corresponding baseline value as covariates. The treatment difference in the least-squares means and the 2-sided 95% CI will be estimated based on this model.

Given the skewed nature of the ACR, the analysis will be performed similarly as described above on the log scale. The percentage of treatment difference, ie, treatment difference in mean ACR relative to placebo, can be calculated by taking the anti-logarithm of the estimated coefficient for the treatment group and subtracting 1. The ratio of mean ACR in treatment compared to placebo and its 95% CI will be presented.

Only subjects with baseline and at least one post-baseline measurement will be included in the analysis. The analysis for proinsulin/insulin ratio will be conducted on subjects who are not receiving insulin at randomization. For subjects who are started on insulin during the study, all proinsulin/insulin data after initiation of insulin will be censored.

Given the skewed nature of the distribution of the percent change in triglycerides, this additional secondary endpoint will be analyzed using nonparametric methods as outlined below. A Wilcoxon rank sum test will be performed. The Hodges-Lehman estimator for the difference in the medians and the distribution-free 95% CIs based on the Wilcoxon rank sum test<sup>3</sup> will also be presented.

The change in these additional secondary endpoints from baseline over time will be explored using an MMRM model similar to the one used to analyze the change in HOMA-B (Section 4.2.2.1).

# 4.3. Multiplicity Adjustment

Per the SAP for the integrated summary, only one alpha is proposed for the testing of the multiple hypotheses based on the integrated data and the data from CANVAS-R alone. The Type I error for these tests will be strictly controlled via a gatekeeping procedure. No alpha is preserved for evaluating hypotheses in CANVAS and all tests will be considered nominal with 2-sided 95% CIs provided for descriptive purposes.

# 4.4. Exploratory Efficacy Endpoints

#### 4.4.1. Definition

The following exploratory endpoints will be analyzed:

• Time to the first occurrence of hospitalization for heart failure;

- Time to the first occurrence of the composite endpoint of hospitalization for heart failure or CV death;
- Time to all-cause mortality;
- Time to the first occurrence of composite endpoint of 40% decrease in eGFR, renal death<sup>a</sup> or requirement for renal replacement therapy;
- Time to the first occurrence of composite endpoint of doubling of SCr, renal death or requirement for renal replacement therapy;
- Time to the first occurrence of composite endpoint of 40% decrease in eGFR, renal death, requirement for renal replacement therapy or CV death;
- Time to the first occurrence of composite endpoint of doubling of SCr, renal death, requirement for renal replacement therapy or CV death;
- Time to the first occurrence of composite endpoint of 40% decrease in eGFR, conversion to macroalbuminuria, renal death or requirement for renal replacement therapy;
- Time to the first occurrence of composite endpoint of doubling of SCr, conversion to macroalbuminuria, renal death or requirement for renal replacement therapy;
- Time to first progression of albuminuria, accompanied by an ACR value increase of greater than or equal to 30% from baseline;
- Time to first regression of albuminuria, accompanied by an ACR value decrease of greater than or equal to 30% from baseline;
- Change in eGFR from baseline to the last off-drug measurement;
- Change in eGFR determined from a between-group comparison of the eGFR slopes using all on-drug measurements of eGFR made from the first on-drug measurement to the final on-drug measurement.

# 4.4.2. Analysis Methods

#### 4.4.2.1. CV Endpoints

The analyses of hospitalization for heart failure and the composite of hospitalization for heart failure or CV death will be based on both the ITT analysis set and the On-Treatment analysis set. The HR of canagliflozin (all canagliflozin group as well as each canagliflozin dose) compared to placebo and its 95% CI will be estimated using a stratified Cox proportional hazards regression model with treatment as the explanatory variable and the history of CV disease (secondary and primary prevention) as the stratification factor.

# 4.4.2.2. All-Cause Mortality

All-cause mortality will be analyzed in both the ITT analysis set and the On-Treatment analysis set using a stratified Cox proportional hazards model with treatment as the explanatory variable and

\_

<sup>&</sup>lt;sup>a</sup> Adjudicated non-CV death with a renal proximate cause is considered as renal death

history of CV disease (secondary and primary prevention) as a stratification factor. The HR of canagliflozin (all canagliflozin group as well as each canagliflozin dose) compared to placebo and its 95% CI will be estimated from the model.

# 4.4.2.3. Renal Endpoints

# 4.4.2.3.1. Composite Endpoints

The components of the renal composite endpoints, such as requirement for renal replacement therapy and doubling of serum creatinine, identified by the investigator or the sponsor for meeting the criteria pre-specified in the charter will be sent to the independent EAC.

The time to the first occurrence of each of the renal composite endpoints (refer to Section 4.4.1) will be analyzed in the ITT analysis set using a Cox proportional hazards model with treatment and baseline eGFR ( $< 60, \ge 60 \text{ mL/min/1.73m}^2$ ) as explanatory variables. The HR of canagliflozin (all canagliflozin as well as each canagliflozin dose) compared to placebo and its 95% CI will be estimated from the model.

#### 4.4.2.3.2. Progression of Albuminuria

For the purpose of an exploratory analysis, progression of albuminuria will be assessed as in Section 4.2.2.2 with the additional condition that it must be accompanied by an increase in ACR value greater than or equal to 30% from baseline. The time to the first occurrence of the event will be analyzed in the ITT analysis set using a Cox proportional hazards regression model with treatment and baseline albuminuria status as the explanatory variables, excluding subjects with baseline macroalbuminuria. The HR of canagliflozin (all canagliflozin as well as each canagliflozin dose) compared to placebo and its 95% CI will be estimated from the model.

### 4.4.2.3.3. Regression of Albuminuria

Regression of albuminuria is defined as at least a one stage improvement of albuminuria, accompanied by an ACR value decrease of greater than or equal to 30% from baseline. The time to the first occurrence of the event will be analyzed in the ITT analysis set, using a Cox proportional hazards regression model with treatment and baseline albuminuria status as the explanatory variables, excluding subjects with baseline normal albuminuria. The HR of canagliflozin (all canagliflozin as well as each canagliflozin dose) compared to placebo and its 95% CI will be estimated from the model.

#### 4.4.2.3.4. eGFR Slope

The time slope of eGFR will be analyzed in the On-Treatment analysis set using a linear mixed effects model with eGFR as a dependent variable, and treatment, baseline eGFR value, time (as a continuous variable), treatment by time interaction as fixed effects, and intercept and time as random effects. The parameter of interest is the coefficient for the treatment-by-time interaction term, which measures the slope difference between canagliflozin and placebo over time. Data will be censored at the date of last study medication plus 2 days.

#### 5. SAFETY

Unless otherwise specified, 2 sets of summaries of AEs will be provided. The first set will be based on the data collected up to 07 January 2014 when INT-6 was first approved. The second set of summaries will focus on the serious AEs and AEs leading to study drug discontinuation throughout the entire study periods.

All other safety analyses and summaries (laboratory tests and vital signs) will be based on data collected throughout the entire study period using either the On-Treatment analysis set or the On-Treatment Pre-INT-6 analysis set, unless otherwise specified.

There will be no imputation of missing values for clinical laboratory test results, vital sign measurements in the safety analyses and there will be no hypothesis testing for results from safety analyses.

The treatment groups will be canagliflozin 100 mg, canagliflozin 300 mg, all canagliflozin, and placebo.

# 5.1. Adjudicated MACE Events

Please refer to Section 4.1 for the primary efficacy analysis of adjudicated MACE events.

#### 5.2. Adverse Events

Adverse events (AEs) will be coded using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA) at the time of database lock.

A treatment-emergent adverse event (TEAE) is defined as an AE with an onset after the initiation of double-blind study medication and before the last study medication date plus 30 days. AEs with a start date prior to initiation of double-blind study medication which are reported to have an increase in intensity, or AEs reported to have an attribution in relationship to study medication (ie, attribution to possible, probably, very likely) after the initiation of double-blind study medication will also be considered as TEAEs. Most of the AE analyses will pertain to the TEAEs.

#### 5.2.1. Adverse Event Collection

As one of the initial studies in the Phase 3 program, CANVAS was designed to collect detailed information on AEs. Upon the approval of canagliflozin in the United States, the safety profile of canagliflozin had been well established. The AE collection was then streamlined following the approval of INT-6 to include only:

- Serious adverse events (SAEs);
- Adverse events that resulted in study drug discontinuation;
- All AEs (serious and non-serious) for AEs of interest (refer to Table 3 below).

For selected AEs of interest, additional data will be collected on supplementary CRF pages primarily for the purposes of narrative description of certain events. Table 3 lists the AEs of interest that will be summarized.

#### **Table 3:** Adverse Events of Interest

Section A. All AEs (serious and non-serious) listed below were collected in CANVAS through INT-6. After INT-6, only the AEs that were serious or that led to study drug discontinuation were collected:

Osmotic diuresis

Volume depletion

Hypoglycemia

Urinary tract infection (UTI)

Female mycotic genital infection

Severe hypersensitivity /cutaneous reactions

**Pancreatitis** 

Hepatic injury

Renal related AEs (including Nephrotoxicity/ acute kidney injury)

# Section B. The AEs listed below were collected regardless of whether they were serious and/or led to study drug discontinuation for the entire study:

Male mycotic genital infection (balanitis, phimosis, events leading to circumcision)

Malignancy

Renal cell cancer

Bladder cancer

Pheochromocytoma

Leydig cell tumors

Breast cancer

Photosensitivity

Venous thromboembolic events (VTE)

Amputation

Fracture

Diabetic ketoacidosis (DKA)

The AEs listed above will be identified using a MedDRA preferred term list (Appendix 1.4).

# 5.2.2. Analysis Methods

The study duration of CANVAS is long relative to the rest of the canagliflozin Phase 3 program. Accordingly, the incidences of AEs (ie, proportion of subjects reporting an AE) reported from this study are not comparable to the incidences generated in the Phase 3 program. Therefore, the exposure-adjusted incidence rate will also be reported in addition to the incidence. The exposure-adjusted incidence rate is calculated as the total number of subjects with the AE divided by the ontreatment exposure in subject-years. For some particular AEs such as malignancy where the off-drug follow up is included, the follow-up-adjusted incidence rate will be estimated. The rate is calculated as the total number of subjects with the related AE divided by the follow-up time in subject-years.

For general AEs and selected AEs of interest that are not routinely collected (refer to Section A of Table 3) after implementation of INT-6, the focus of the summary will be the serious AEs and the AEs leading to discontinuation of study medication.

#### 5.2.2.1. General Adverse Events

#### **Prior to the Approval of INT-6**

On-Treatment Pre-INT6 analysis set will be used for the summary of general AEs prior to the approval of INT-6 unless otherwise specified.

The overall incidence and the exposure-adjusted incidence rate of AEs, AEs leading to discontinuation, drug-related AEs, drug-related AEs leading to discontinuation, SAEs, SAEs leading to discontinuation, serious drug-related AEs, serious drug-related AEs leading to discontinuation, and deaths will be summarized by treatment group.

AEs by System Organ Class (SOC) will be summarized by treatment group.

For each AE, the percentage of subjects who experienced at least one occurrence of the given event will be provided by preferred term, grouped by SOC, and presented by treatment group. In addition, the incidence of severe AEs and drug-related AEs (possibly related, probably related and very likely related, as reported by the investigator) will be summarized by preferred term, grouped by SOC, and presented by treatment group). The incidence of AEs (by preferred term, grouped by SOC, and presented by treatment group) will also be summarized by the action taken regarding the study medication, as well as by the outcome.

For reference, as a screening tool, the 95% CIs for incidence difference between treatment groups will be calculated for the AEs which are reported in at least 4 subjects in any treatment group. Four (rule-of-4) was chosen based on the recommendation from the Safety, Planning, Evaluation, and Reporting Team (SPERT).<sup>4</sup> The exclusion of "0" from the 95% CI for the between-group difference in incidence for a particular AE does not necessarily imply that the difference is due to the drug. The intent of providing the 95% CIs is as a filter to identify AEs that require additional assessment. AEs identified by the above screening procedure will be presented and subject to further evaluation.

#### **Through the Entire Study**

Serious AEs and the AEs leading to discontinuation collected throughout the entire study will be analyzed based on On-Treatment analysis set unless otherwise specified.

An overview summary table with the incidence and the exposure-adjusted incidence will be generated for:

- Serious AEs;
- Deaths;
- AEs leading to discontinuation of study medication;
- Serious AEs leading to discontinuation of study medication;
- Serious AEs considered drug-related;
- AEs considered drug-related leading to discontinuation of study medication.

SAEs by SOC and preferred term will be summarized by treatment group using the On-Treatment analysis set. The same summary will be provided for AEs leading to discontinuation of study medication using the On-Treatment analysis set.

The incidence of all SAEs (by preferred term, grouped by SOC, and presented by treatment group) will also be summarized by the relationship to study drug, by the action taken regarding the study drug, as well as by the outcome. The relationship to study drug will be presented by 2 categories: related (which includes possibly related, probably related and very likely related, as reported by the investigator) and not related (which includes not related and doubtfully related, as reported by the investigator).

For reference, as a screening tool, the 95% CIs for incidence difference between treatment groups will be calculated for the AEs (regardless of seriousness) which are reported in at least 4 or more subjects in any treatment group. Only the AEs identified by the above screening procedure will be presented and subject to further evaluation.

Listings will also be provided for deaths, SAEs, and AEs leading to study drug discontinuation.

For AEs of interest in Section A of Table 3 (with the exception of hypoglycemia, see Section 5.2.2.3), a summary similar to the analysis of general AEs will be provided. The AEs will be identified using the MedDRA preferred terms listed in Appendix 1.4.

#### **5.2.2.2.** Male Mycotic Genital Infections

Balanitis and phimosis AEs will be identified using the MedDRA preferred terms listed in Appendix 1.4 and the analyses will be based on On-Treatment analysis set only.

Using the On-Treatment analysis set, an overview summary table with the incidence and the exposure-adjusted incidence will be provided for:

- All AEs;
- Serious AEs:
- AEs considered drug-related AEs leading to discontinuation of study medication;
- Serious AEs leading to discontinuation of study medication;
- Serious AEs considered drug-related;
- AEs considered drug-related leading to discontinuation of study medication.

AEs by preferred term will be summarized by treatment group. A Kaplan-Meier plot for the time to first occurrence of balanitis will be provided by treatment group.

In addition, circumcision events will be identified based on blinded medical review of the clinical database prior to the database lock and summarized by treatment group.

Based on the additional information collected on the designated supplemental eCRF page in CANVAS, the following additional study-specific analyses will be performed:

- The incidence of male subjects with any genital mycotic infections will be summarized by treatment group and by circumcision status.
- Descriptive statistics (N, mean, SD, median, and range) will be calculated by treatment group for the duration (days) and severity (grouped as mild or moderate vs. severe) of all infections. If a subject experienced multiple events, all durations will be included in the summary.
- Descriptive statistics (N, mean, SD, median, and range) will be calculated by treatment group for the number of days from start of the AE treatment to the resolution of the symptoms.

## 5.2.2.3. Hypoglycemia

Hypoglycemia episodes were collected by a specific, dedicated eCRF for all hypoglycemia up to INT-6. Hypoglycemia episodes reported on the supplemental eCRF up to 07 January 2014 will be analyzed based on On-Treatment Pre-INT6 analysis set. For hypoglycemia reported on the general AE page throughout the study period, focus will be the serious events or the events leading to study drug discontinuation.

# **Prior to the Approval of INT-6**

A subject will be counted as having a documented hypoglycemia episode when there is either a biochemically documented hypoglycemic episode (ie, concurrent fingerstick glucose or plasma glucose  $\leq 70 \text{ mg/dL}$  [3.9 mmol/L]), and/or a severe hypoglycemic episode as reported on the hypoglycemia eCRF, as follows:

- Biochemically documented hypoglycemia episode: a hypoglycemia episode with a concurrent reported glucose value of  $\leq 70 \text{ mg/dL}$  (3.9 mmol/L), regardless of whether the episode is associated with symptoms (symptomatic hypoglycemia) or not (asymptomatic hypoglycemia).
- Severe hypoglycemia episode: a hypoglycemia episode that has the answer "Yes" recorded for any of the following 3 questions on the hypoglycemia eCRF: "Did the subject require the assistance of others to treat?", "Did the subject lose consciousness during the episode?", or "Did the subject have a seizure during the episode?"

Only treatment emergent hypoglycemia episodes, reported on the eCRF for hypoglycemia, will be summarized. Treatment emergent is defined the same way as TEAEs (defined in Section 5.2).

The percentages of subjects with documented hypoglycemia episodes (ie, biochemically documented and/or severe) and subjects with biochemically documented, and with severe hypoglycemia episodes separately, will be summarized by treatment group. For subjects with biochemically documented hypoglycemia episodes, the percentage of subjects will be summarized for each of the following glucose levels (≤70 mg/dL [3.9 mmol/L], <56 mg/dL [3.1 mmol/L], and <36 mg/dL [2.0 mmol/L], "Low" results will be included in all 3 categories) by treatment group. For subjects with severe hypoglycemia episodes, the percentage of subjects by each answer of the 3 questions for severe hypoglycemia on the eCRF will be summarized by treatment group. The

event rate by person-year (total number of episodes/total exposure) will be calculated by treatment group separately for documented and for severe hypoglycemia.

Subjects who had 0, 1, 2, or  $\ge 3$  documented episodes and subjects who had 0, 1, 2, or  $\ge 3$  severe hypoglycemic episodes will be summarized by treatment group.

In addition, the incidence of all episodes of hypoglycemia reported on the eCRF for hypoglycemia will be summarized (this includes events without concurrent fingerstick glucose reported and events with fingerstick glucose > 70 mg/dL [3.9 mmol/L]) by treatment group.

# **Through the Entire Study**

Using the On-Treatment analysis set, an overview summary table with the incidence and the exposure-adjusted incidence will be provided for:

- Serious AEs;
- AEs leading to discontinuation of study medication;
- Serious AEs leading to discontinuation of study medication;
- Serious AEs considered drug-related;
- AEs considered drug-related leading to discontinuation of study medication;

SAEs by preferred term will be summarized by treatment group.

# 5.2.2.4. Selected Malignancies

The selected malignancies of interest are renal cell cancer, bladder cancer, testicular cancer (Leydig cell tumors), pheochromocytomas, and breast cancer. Selected malignancy AEs will be identified using the MedDRA preferred terms listed in Appendix 1.4 and the analyses will be based on the On-Study analysis set.

For each selected malignancy of interest, an overview summary table with the incidence and the follow-up-adjusted incidence will be provided for:

- All AEs:
- Serious AEs;
- AEs considered drug-related (investigator assessment of possible, probable or very likely);
- AEs leading to discontinuation of study medication;
- Serious AEs leading to discontinuation of study medication;
- Serious AEs considered drug-related;
- AEs considered drug-related leading to discontinuation of study medication.

The preferred terms associated with each selected malignancy type will be summarized by treatment.

# 5.2.2.5. Photosensitivity

Photosensitivity AE will be identified using the MedDRA preferred terms listed in Appendix 1.4 and the analyses will use the On-Treatment analysis set.

An overview summary table with the incidence and the exposure-adjusted incidence will be provided for:

- All AEs;
- Serious AEs;
- AEs considered drug-related (investigator assessment of possible, probable or very likely);
- AEs leading to discontinuation of study medication;
- Serious AEs leading to discontinuation of study medication;
- Serious AEs considered drug-related;
- AEs considered drug-related leading to discontinuation of study medication.

AEs by preferred term will be summarized by treatment group.

#### 5.2.2.6. Venous Thromboembolic Events

Venous thromboembolic (VTE) events will be identified using the list of MedDRA terms in Appendix 1.4. Adverse events identified by the investigator or the sponsor for meeting the criteria pre-specified in the charter will be sent to the independent EAC for confirmation. The analyses will use the On-Treatment analysis set of adjudicated VTEs. Additionally, a similar analysis of investigator reported VTE events will also be provided.

An overview summary table with the incidence and the exposure-adjusted incidence will be provided for:

- All AEs;
- Serious AEs;
- AEs considered drug-related (investigator assessment of possible, probable or very likely);
- AEs leading to discontinuation of study medication;
- Serious AEs leading to discontinuation of study medication;
- Serious AEs considered drug-related;
- AEs considered drug-related leading to discontinuation of study medication.

AEs by preferred term will be summarized by treatment group.

The incidence of VTEs identified by the MedDRA preferred terms listed in Appendix 1.4 will also be summarized by preferred term. A summary table of all VTEs (regardless of adjudication) will also be provided by preferred term.

#### **5.2.2.7.** Fracture

Fracture events identified by the investigator or the sponsor for meeting the criteria pre-specified in the charter will be sent to the independent Fracture Adjudication Committee to confirm that events were fractures, to determine fracture location (anatomic region) and type (low trauma or not). The main analysis will be based on the adjudicated low trauma fractures in the On-Study analysis set.

An overview summary table with the incidence and the follow-up-adjusted incidence will be provided for:

- Adjudicated fractures;
- Adjudicated fractures considered serious (investigator assessment);
- Adjudicated fractures considered drug-related (investigator assessment of possible, probable or very likely);
- Adjudicated fractures leading to discontinuation of study medication;
- Adjudicated fractures considered serious and drug-related (investigator assessment);
- Adjudicated fractures considered drug-related (investigator assessment) and leading to discontinuation of study medication.

A summary of adjudicated fracture stratified by anatomical region by treatment will be provided. The incidence as well as the incidence rate will be presented.

A Kaplan-Meier plot for the time to the first occurrence of adjudicated fracture event will be provided by treatment group. The HR and the 95% CI will be derived from a Cox proportion hazards model with a term for treatment as an explanatory variable. The HR will be estimated in subgroups based on sex, baseline age (<65 and  $\ge65$  years), duration of T2DM (<10 and  $\ge10$  years), baseline eGFR (<60 and  $\ge60$  mL/min/1.73 m<sup>2</sup>), and prior fracture history (yes or no).

A summary of all adjudicated fractures by anatomic location will be provided. The HR and its 95% CI as well as a Kaplan-Meier plot for the first occurrence of all adjudicated fractures will be provided using the same analysis as low trauma fracture.

# 5.2.2.8. Amputation

The main analysis of lower extremity amputations as documented in the dedicated eCRF will be based on the On-Study analysis set. An overview summary table with the incidence and the follow-up-adjusted incidence will be provided for:

- All lower limb amputations;
- Traumatic lower limb amputation;
- Atraumatic lower limb amputation.

Summary of anatomical region (toe, ankle, trans-metatarsal, below knee, above knee) of lower extremity atraumatic amputations will be reported by treatment group.

For atraumatic lower limb amputation, a Kaplan-Meier plot for the time to the first occurrence of event will be provided by treatment group. The association of amputation with treatment and the baseline risk factors listed in Table 4 will be assessed via logistic regression modeling. The relationship between amputation and some post-treatment factors such as volume depletion will also be explored.

For the post-treatment AEs that may be associated with amputation, groupings of selected MedDRA preferred terms used to identify events to be included in each of the following SOC categories are presented in Appendix 1.5:

- Infections and Infestations:
- Vascular disorders;
- Nervous System disorders;
- Skin and subcutaneous tissue disorders;
- Osteomyelitis.

The selected preferred terms in infections and infestation are further split into "Reversible Infection" and "Irreversible Infections". In addition, the preferred terms grouped under the MedDRA high level term of "skin and subcutaneous tissue ulcerations" are also of interest.

For each AE group listed above, the incidence of the respective preferred terms will be summarized by treatment. Stratified by treatment, the odds ratio of amputation and each AE group listed above will be estimated.

**Baseline Factors Included in the Logistic Regression Analysis** 

| Gender | <ul> <li>Smoking</li> </ul> |
|---|---|
| <ul> <li>Cardiovascular disease history</li> </ul> | • Use of insulin |
| Peripheral vascular disease history <sup>a</sup> | <ul> <li>Baseline Systolic Blood Pressure</li> </ul> |
| <ul> <li>Amputation history</li> </ul> | $\circ$ > 120 vs $\leq$ 120 mmHg |
| <ul> <li>Neuropathy history</li> </ul> | $\circ > 140 \text{ vs } \leq 140 \text{ mmHg}$ |
| <ul> <li>Retinopathy history</li> </ul> | • Baseline eGFR (ml/min/1.73m <sup>2</sup> ) |
| <ul> <li>Nephropathy history</li> </ul> | $\circ$ < 60 vs $\geq$ 60 |
| Any diuretic use | o < 45 vs ≥45 |
| Loop diuretic use | • Diabetes duration (< 10 vs ≥10 yrs.) |
| Non-loop diuretic use | • Baseline $HbA_{1c}$ (> 8 vs $\leq$ 8%) |

 $eGFR (mL/min/1.73m^2)$ Age (yrs.) Diabetes duration (yrs.) HbA<sub>1c</sub> (%) Systolic blood pressure (mmHg) Hemoglobin (g/L)

Excludes amputation history

#### 5.2.2.9. Diabetic Ketoacidosis

Diabetic ketoacidosis (DKA) and related AEs will be identified using the list of MedDRA terms in Appendix 1.4. Adverse events identified by the investigator or the sponsor for meeting the criteria pre-specified in the charter will be sent to the independent DKA Adjudication Committee. The main analysis of the DKA events will be based on adjudicated events of DKA in the On-Study analysis set. Events occurring at any time post-randomization, regardless of the timing of the last dose of study medication, will be included.

For the adjudicated DKA events, a table will summarize the incidence and the follow-up-adjusted incidence rate.

A listing of all DKA events identified by the sponsor's medical monitoring team and the subset of the events that went for adjudication will be provided.

#### 5.2.2.10. Pancreatitis

Pancreatitis and related AEs identified by the sponsor using the list of MedDRA terms prespecified in the charter will be sent to the independent Pancreatitis Adjudication Committee. The main analysis of events will be based on adjudicated, confirmed events in the On-Treatment analysis set. Analysis based on events occurring at any time post-randomization, regardless of the timing of the last dose of study medication, will be performed. The incidence rate and proportion of adjudicated pancreatitis events by severity will be summarized. The total number of subjects with an event not confirmed by the Pancreatitis Adjudication Committee will also be summarized.

# 5.3. Clinical Laboratory Tests

A list of clinical laboratory assessments made during the study is provided in Appendix 1.2. The percentage of subjects with specific treatment-emergent laboratory values meeting pre-defined limit of change (PDLC) criteria listed in Appendix 1.3 will be summarized. The 95% CI for the percentage difference between canagliflozin compared to the placebo group will be provided for each PDLC criterion which has at least 4 or more subjects in any treatment group. A corresponding listing will also be provided. As described above, PDLC values will be presented based on measurements on study drug, and up to a maximum of 2 days after the last dose of study drug, as well as all measurements regardless of the time of the last dose of double-blind study drug. Summaries based on both standard units (SI) and conventional units will be provided.

# 5.4. Vital Signs

A treatment-emergent vital sign abnormality is defined as a change from baseline and subsequent post-baseline value that satisfies the PDLC criteria listed in Appendix 1.3. For each vital sign parameter, the proportion of subjects with a treatment-emergent abnormality will be tabulated by treatment group. PDLC values will be presented based on measurements up to a maximum of 2 days after the last dose of study drug.

The blood pressure measurements will be based on the average of the consecutive sitting blood pressure readings that were to be collected at each visit.

# 5.5. Electrocardiogram

The decision was made to stop collecting ECG measurements after Week 52 since INT-6. The analyses will use all the ECG data available up to the approval of INT-6. The ECG variables that will be analyzed are heart rate, PR interval, QRS interval, QT interval, and QTc using the Fridericia (QTcF) correction methods. The QTcF corrected interval values are based on the following formula:<sup>5</sup>

• Fridericia: QTcF (msec) = QT(msec) \* (HR(bpm)/60)1/3.

The PDLC criteria for defining an ECG abnormality for PR interval, QRS interval, QTcF values, and changes from baseline within each category are listed in Appendix 1.3. The number and the percentage of subjects in each category will be summarized by treatment group up to 2 days after the last dose of study drug.

# **REFERENCES**

- 1. Little R et al. The treatment of missing data in a large cardiovascular clinical outcomes study. *Clin Trials*. 2016;13(3):344-51.
- 2. KDOQI 2007. National Kidney Foundation Kidney Disease Outcomes Quality Initiative (KDOQI). *Amer J of Kidney Diseases* 2007;49(2, Suppl 2):S1-S180.
- 3. Hollander M, Wolfe DA. Nonparametric Statistical Methods, Second edition. John Wiley and Sons, Inc., 1999.
- 4. Crowe BJ, Xia HA, Berlin JA, et al. Recommendations for safety planning, data collection, evaluation and reporting during drug, biologic and vaccine development: a report of the safety planning, evaluation, and reporting team. *Clin Trials*. 2009;6:430-440.
- 5. Fridericia LS. The duration of systole in the electrocardiogram of normal subjects and of patients with heart disease. *Acta Medica Scandinavica*. 1920; 53:469 486.

Approved, Date: 20 March 2017
## **APPENDIX**

## Appendix 1.1: List of Key Analyses of CV and Mortality Endpoints

| Analysis Set | Endpoint | Section |
|---|---|---|
| Primary Efficacy As | ssessment of MACE | |
| ITT | MACE | 4.1.2 |
| On-Study | MACE | 4.1.4.1 |
| On-Treatment | MACE | 4.1.4.2 |
| ITT | MACE components | 4.1 |
| On-Treatment | MACE components | 4.1 |
| ITT | Subgroup analysis of MACE | 4.1.3 |
| Exploratory Assessn | nent of Additional CV Endpoints | |
| ITT | Hospitalization for heart failure | 4.4.2.1 |
| On-Treatment | Hospitalization for heart failure | 4.4.2.1 |
| ITT | Composite of hospitalization for heart failure or CV Death | 4.4.2.1 |
| On-Treatment | Composite of hospitalization for heart failure or CV Death | 4.4.2.1 |
| ITT | All-cause Mortality | 4.4.2.2 |

### **Appendix 1.2: Clinical Laboratory Tests**

The clinical laboratory tests include following panels and assessments:

- Hematology panel
  - hemoglobin
  - o platelet count
  - hematocrit
  - o red blood cell (RBC) count
  - o white blood cell (WBC) count with differential
- Serum chemistry panel

 Sodium o alkaline phosphatase o creatine phosphokinase (CPK) o potassium lactic acid dehydrogenase (LDH) o chloride o bicarbonate o uric acid o BUN o calcium o creatinine o phosphate o albumin o aspartate aminotransferase (AST) o alanine aminotransferase (ALT) o total protein o gamma-glutamyltransferase (GGT) o magnesium

- total bilirubin
- Fasting serum lipid profile (triglycerides, LDL-C, HDL-C, total cholesterol).
- HbA<sub>1c</sub>
- Urinalysis (dipstick analysis; from spot urine collection in the clinic on Day 1; performed at central laboratory; microscopic analysis is not required). Urine glucose will not be measured by the central laboratory.
  - o specific gravity ketones
  - o pH bilirubin/urobilinogen
  - o protein nitrite
  - blood leukocyte esterase
- Central laboratory will report the estimated glomerular filtration rate (eGFR) according to the Modification of Diet in Renal Disease Study (MDRD) equation (Levey 2006) at study visits when serum creatinine is measured. The 4-variable MDRD eGFR includes serum creatinine, age, race, and sex according to the equation below:

For creatinine in mg/dL:

```
eGFR (mL/min/1.73 m<sup>2</sup>) = 175 x (serum creatinine) ^{-1.154} x (age) ^{-0.203} x (0.742 if female) x (1.21 if black)
```

For creatinine in µmol/L:

eGFR (mL/min/1.73m<sup>2</sup>) = 175 x (serum creatinine x 0.0113)  $^{-1.154}$  x (age)  $^{-0.203}$  x (0.742 if female) x (1.21 if black)

# Appendix 1.3: Pre-defined Limit of Change (PDLC) Criteria

| <b>Laboratory Test</b> | Parameter for ANY value and LAST value |
|---|---|
| CHEMISTRY | |
| Albumin | Composite: <lln and="">25% decrease from BL</lln> |
| Absolute Value: >3X ULN | |
| ALT | Absolute Value: >5X ULN |
| | Absolute Value: >8X ULN |
| | Absolute Value: >3X ULN |
| AST | Absolute Value: >5X ULN |
| | Absolute Value: >8X ULN |
| | Composite: ALT >3X ULN and Tbili >2X ULN [with the Tbili elevation >2 |
| ALT >3X ULN and Tbili >2X ULN | X ULN within 30 days of the ALT elevation >3x ULN] |
| | Composite: AST >3X ULN and Tbili >2X ULN [with the Tbili elevation >2 X |
| AST >3X ULN and Tbili >2X ULN | ULN within 30 days of the AST elevation >3x ULN] |
| | Composite: >ULN and > 25% increase from BL |
| Bilirubin | Absolute Value: >2XULN |
| Bicarbonate | Absolute Value: <16 mEq/L |
| Calcium | Composite: >ULN and > 10 % increase from BL |
| Creatinine Kinase | Absolute Value: >1000U/L |
| | Composite: < 80 and decrease>30% from BL |
| eGFR | Change: decrease>50% from BL |
| | Composite: <lln and="">25% decrease from BL</lln> |
| Magnesium | Composite: >ULN and >25% increase from BL |
| Phosphorus | Composite: >ULN and >25% increase from BL |
| | Composite: <lln and="">15% decrease from BL</lln> |
| Potassium | Composite: >ULN and >15% increase from BL |
| | Absolute Value: ≥ 6.5 mEq/L |
| | Composite: <lln and="" decrease="">5 mEq/L or more from BL</lln> |
| Sodium | Composite: >ULN and increase>5 mEq/L or more from BL |
| Uric Acid | Composite: <lln and="">25% decrease from BL</lln> |
| HEMATOLOGY | |
| | Change: ≥ 2 g/dl decrease from BL |
| Hemoglobin | Change: ≥ 2 g/dL increase from BL |
| Platelets | Composite: >ULN and increase >25% from BL |
| | Composite: < LLN and >25% decrease from BL |
| White Blood Count | Composite: > ULN and >50 % increase from BL |
| VITAL SIGNS | |
| | Absolute Value: ≤50 beats per minute |
| Pulse | Absolute Value: ≥100 beats per minute |
| | Composite: ≥ 20 mm Hg decrease from BL and ≤90 mm Hg |
| Systolic Blood Pressure | Composite: ≥ 20 mm Hg increase from BL and ≥ 160 mm Hg |
| | Composite: ≥ 15 mm Hg decrease from BL and ≤ 50 mm Hg |
| Diastolic Blood Pressure | Composite: ≥ 15 mm Hg increase from BL and ≥ 100 mm Hg |
| ECG PARAMETERS | |
| | Change: >30-60 ms |
| | Change: >60 ms |
| QTcF | |
| | Absolute Value: > 450-480 ms |
| | Absolute Value: > 480-500 ms |
| | Absolute Value: >500 ms |
| PR Interval | Absolute Value: ≥ 200 ms |
| QRS Interval | Absolute Value: ≤ 50 ms |
| AV2 IIIci vai | Absolute Value: ≥ 120 ms |

39

## Appendix 1.4: List of Preferred Terms for Selected AEs of Interest

| | Famala Massatia Carital | |
|---|---|---|
| Diabetic ketoacidosis | Female Mycotic Genital Infections | Fracture |
| Acidosis | Genital candidiasis | Acetabulum fracture |
| Acidosis aggravated | Genital infection | Ankle fracture |
| Acidosis diabetic | Genital infection female | Atypical femur fracture |
| Acidosis metabolic | Genital infection fungal | Atypical fracture |
| Acidosis NOS | Urogenital infection fungal | Avulsion fracture |
| Acute acidosis | Vaginal infection | Bone fragmentation |
| Anion gap acidosis | Vaginal inflammation | Cervical vertebral fracture |
| Blood ketone body | Vulvitis | Chance fracture |
| Blood ketone body increased | Vulvovaginal candidiasis | Clavicle fracture |
| | Vulvovaginal mycotic | |
| Blood ketone body present | infection | Closed fracture manipulation |
| Diabetes mellitus with ketoacidosis | Vulvovaginitis | Comminuted fracture |
| Diabetes with hyperosmolarity | č | Complicated fracture |
| Diabetes with ketoacidosis | | Compression fracture |
| Diabetic acidosis | | Craniofacial fracture |
| Diabetic hyperglycemic coma | | Elevation skull fracture |
| Diabetic hyperosmolar coma | | Epiphyseal fracture |
| Diabetic ketoacidosis | | External fixation of fracture |
| Diabetic ketoacidotic hyperglycemic | | |
| coma | | Facial bones fracture |
| Diabetic metabolic decompensation | | Femoral neck fracture |
| High anion gap metabolic acidosis | | Femur fracture |
| Hyperglycemic seizure | | Fibula fracture |
| Hyperosmolar hyperglycemic state | | Foot fracture |
| Hyperosmolar state | | Forearm fracture |
| Ketoacidosis | | Fracture |
| Ketonuria | | Fracture debridement |
| Ketosis | | Fracture delayed union |
| Metabolic acidosis | | Fracture displacement |
| Metabolic acidosis exacerbated | | Fracture malunion |
| Metabolic acidosis NOS exacerbated | | Fracture nonunion |
| Metabolic acidosis not otherwise | | F |
| specified (NOS) | | Fracture pain |
| Metabolic acidosis worsened | | Fracture reduction |
| Type I diabetes mellitus with ketoacidosis | | Enochana traceture and |
| | | Fracture treatment |
| Type II diabetes mellitus with ketoacidosis | | Fractured coccyx |
| Retoactuosis | | Fractured coccyx Fractured ischium |
| | | Fractured ischium Fractured maxilla elevation |
| | | Fractured sacrum |
| | | Fractured skull depressed |
| | | Fractured zygomatic arch elevation |
| | | Greenstick fracture |
| | | Hand fracture |
| | | Hip fracture |
| | | Humerus fracture |
| | | Ilium fracture |
| | | Impacted fracture |
| | | Internal fixation of fracture |
| | | Jaw fracture |
| | | Limb crushing injury |
| | | Limb fracture |

| | Female Mycotic Genital | |
|---|---|---|
| Diabetic ketoacidosis | Infections | Fracture |
| | | Loss of anatomical alignment after fracture |
| | | reduction |
| | | Lower limb fracture |
| | | Lumbar vertebral fracture |
| | | Multiple fractures |
| | | Open fracture |
| | | Open reduction of fracture |
| | | Open reduction of spinal fracture |
| | | Osteochondral fracture |
| | | Osteoporotic fracture |
| | | Patella fracture |
| | | Pathological fracture |
| | | Pelvic fracture |
| | | Periprosthetic fracture |
| | | Pubis fracture |
| | | Radius fracture |
| | | Rib fracture |
| | | Sacroiliac fracture |
| | | Scapula fracture |
| | | Skull fracture |
| | | Skull fractured base |
| | | Spinal compression fracture |
| | | Spinal fracture |
| | | Spinal fusion fracture |
| | | Sternal fracture |
| | | Stress fracture |
| | | Thoracic vertebral fracture |
| | | Tibia fracture |
| | | Torus fracture |
| | | Traumatic fracture |
| | | Ulna fracture |
| | | Upper limb fracture |
| | | Wrist fracture |

| Hepatic Injury | Hypoglycaemia | Male Mycotic Genital Infections |
|---|---|---|
| Acute graft versus host disease in liver | Hypoglycaemia | Balanitis |
| Acute hepatic failure | Hypoglycaemic coma | Balanitis candida |
| Acute yellow liver atrophy | Hypoglycaemic seizure | Balanoposthitis |
| Allergic hepatitis | | Balanoposthitis infective |
| Ammonia increased | | Erosive balanitis |
| Ascites | | Gangrenous balanitis |
| Asterixis | | Genital candidiasis |
| Autoimmune hepatitis | | Genital infection |
| Bacterascites | | Genital infection fungal |
| Biliary ascites | | Genital infection male |
| Biliary cirrhosis | | Penile infection |
| Biliary cirrhosis primary | | Posthitis |
| Biliary fibrosis | | |
| Bilirubin excretion disorder | | |
| Biopsy liver abnormal | | |
| Child-Pugh-Turcotte score increased | | |
| Cholaemia | | |
| Cholestasis | | |
| Cholestatic liver injury | | |
| Cholestatic pruritus | | |
| | | 41 |

#### **Hepatic Injury**

#### Hypoglycaemia

#### **Male Mycotic Genital Infections**

Chronic graft versus host disease in

liver

Chronic hepatic failure

Chronic hepatitis

Coma hepatic

Cryptogenic cirrhosis

Diabetic hepatopathy

Drug-induced liver injury

Duodenal varices

Focal nodular hyperplasia

Gallbladder varices

Gastric varices

Gastric varices haemorrhage

Graft versus host disease in liver

Haemangioma of liver

Haemorrhagic ascites

Haemorrhagic hepatic cyst

Hepatectomy

Hepatic adenoma

Hepatic atrophy

Hepatic calcification

Hepatic cirrhosis

Hepatic cyst

Hepatic cyst ruptured

Hepatic encelalopathy

Hepatic encephalopathy prophylaxis

Hepatic failure

Hepatic fibrosis

Hepatic fibrosis marker abnormal

Hepatic haemangioma rupture

Hepatic hydrothorax

Hepatic infiltration eosinophilic

Hepatic lesion

Hepatic necrosis

Hepatic steatosis

**Hepatitis** 

Hepatitis acute

Hepatitis cholestatic

Hepatitis chronic active

Hepatitis chronic persistent

Hepatitis fulminant

Hepatitis toxic

Hepatobiliary disease

Hepatocellular foamy cell syndrome

Hepatocellular injury

Hepatopulmonary syndrome

Hepatorenal failure

Hepatorenal syndrome

Hepatotoxicity

Hyperbilirubinaemia

Icterus index increased

Intestinal varices

Ischaemic hepatitis

Jaundice

Jaundice cholestatic

Jaundice hepatocellular

Liver and small intestine transplant

| Hepatic Injury | Hypoglycaemia | Male Mycotic Genital Infections |
|---|---|---|
| Liver disorder | | |
| Liver injury | | |
| Lupoid hepatic cirrhosis | | |
| Lupus hepatitis | | |
| Mixed liver injury | | |
| Nodular regenerative hyperplasia | | |
| Non-alcoholic steatohepatitis | | |
| Non-cirrhotic portal hypertension | | |
| Ocular icterus | | |
| Oedema due to hepatic disease | | |
| Oesophageal varices haemorrhage | | |
| Parenteral nutrition associated liver | | |
| disease | | |
| Peripancreatic varices | | |
| Periportal oedema | | |
| Portal hypertension | | |
| Portal hypertensive enteropathy | | |
| Portal hypertensive gastropathy | | |
| Portal triaditis | | |
| Portal vein cavernous transformation | | |
| Portal vein dilatation | | |
| Portopulmonary hypertension | | |
| Radiation hepatitis | | |
| Renal and liver transplant | | |
| Retrograde portal vein flow | | |
| Reye's syndrome | | |
| Reynold's syndrome | | |
| Splenic varices | | |
| Splenic varices haemorrhage | | |
| Subacute hepatic failure | | |
| Varices oesophageal | | |
| Varicose veins of abdominal wall | | |

| Malignancy Bladder Cancer | Malignancy Breast Cancer | Malignancy Phaeochromocytoma |
|---|---|---|
| Bladder adenocarcinoma recurrent | Apocrine breast carcinoma | Phaeochromocytoma |
| Bladder adenocarcinoma stage 0 | Breast angiosarcoma | Phaeochromocytoma crisis |
| • | Breast angiosarcoma | • |
| Bladder adenocarcinoma stage I | metastatic | Phaeochromocytoma excision |
| Bladder adenocarcinoma stage II | Breast cancer | Phaeochromocytoma malignant |
| Bladder adenocarcinoma stage III | Breast cancer female | |
| Bladder adenocarcinoma stage IV | Breast cancer in situ | |
| Bladder adenocarcinoma stage unspecified | Breast cancer male | |
| Bladder cancer | Breast cancer metastatic | |
| Bladder cancer recurrent | Breast cancer recurrent | |
| Bladder cancer stage 0, with cancer in situ | Breast cancer stage I | |
| Bladder cancer stage 0, without cancer in | | |
| situ | Breast cancer stage II | |
| Bladder cancer stage I, with cancer in situ | Breast cancer stage III | |
| Bladder cancer stage I, without cancer in | | |
| situ | Breast cancer stage IV | |
| Bladder cancer stage II | Breast neoplasm | |
| Bladder cancer stage III | Breast sarcoma | |
| Bladder cancer stage IV | Breast sarcoma metastatic | |
| Bladder squamous cell carcinoma recurrent | Breast sarcoma recurrent | |
| Bladder squamous cell carcinoma stage 0 | Contralateral breast cancer | |
| - | | |

| Malignancy Bladder Cancer | Malignancy Breast Cancer | Malignancy Phaeochromocytoma |
|---|---|---|
| Bladder squamous cell carcinoma stage I | HER-2 positive breast cancer | |
| | Hormone refractory breast | |
| Bladder squamous cell carcinoma stage II | cancer | |
| | Inflammatory carcinoma of | |
| Bladder squamous cell carcinoma stage III | breast recurrent | |
| | Inflammatory carcinoma of | |
| Bladder squamous cell carcinoma stage IV | breast stage III | |
| Bladder squamous cell carcinoma stage | Inflammatory carcinoma of | |
| unspecified | breast stage IV | |
| | Inflammatory carcinoma of | |
| Bladder transitional cell carcinoma | the breast | |
| Bladder transitional cell carcinoma | Intraductal papillary breast | |
| metastatic | neoplasm | |
| Bladder transitional cell carcinoma | Intraductal proliferative breast | |
| recurrent | lesion Invasive breast carcinoma | |
| Bladder transitional cell carcinoma stage 0 | | |
| Dladder transitional call carainama stage I | Invasive ductal breast carcinoma | |
| Bladder transitional cell carcinoma stage I | Invasive lobular breast | |
| Bladder transitional cell carcinoma stage II | carcinoma | |
| Bladder transitional cell carcinoma stage | Invasive papillary breast | |
| III | carcinoma | |
| Bladder transitional cell carcinoma stage | Lobular breast carcinoma in | |
| IV | situ | |
| Metastases to bladder | Malignant nipple neoplasm | |
| | Malignant nipple neoplasm | |
| Metastatic carcinoma of the bladder | female | |
| | Malignant nipple neoplasm | |
| Transitional cell carcinoma | male | |
| | Medullary carcinoma of breast | |
| | Metaplastic breast carcinoma | |
| | Metastases to breast | |
| | Mucinous breast carcinoma | |
| | Neuroendocrine breast tumour | |
| | Nipple neoplasm | |
| | Oestrogen receptor positive | |
| | breast cancer | |
| | Paget's disease of nipple | |
| | Phyllodes tumour | |
| | Triple negative breast cancer | |
| | Tubular breast carcinoma | |

| Malignancy Renal Cell Cancer | Malignancy Testicular | Osmotic Diuresis |
|---|---|---|
| Clear cell renal cell carcinoma | Benign neoplasm of testis | Dry mouth |
| Clear cell sarcoma of the kidney | Leydig cell tumour of the testis | Dry throat |
| Denys-Drash syndrome | Sertoli cell testicular tumour | Micturition disorder |
| Hereditary leiomyomatosis renal cell carcinoma | Spermatocytic seminoma | Micturition urgency |
| Hereditary papillary renal carcinoma | Testicle adenoma | Nocturia |
| Metastatic renal cell carcinoma | Testicular cancer metastatic | Pollakiuria |
| Nephroblastoma | Testicular neoplasm | Polydipsia |
| Non-renal cell carcinoma of kidney | Testicular papilloma | Polyuria |
| Renal cancer | Testis cancer | Thirst |
| Renal cancer metastatic | | Tongue dry |
| Renal cancer recurrent | | Urine output increased |
| Renal cancer stage I | | • |
| Renal cancer stage II | | |
| Renal cancer stage III | | |
| Renal cancer stage IV | | |
| Renal cell carcinoma | | |
| Renal cell carcinoma recurrent | | |
| Renal cell carcinoma stage I | | |
| Renal cell carcinoma stage II | | |
| Renal cell carcinoma stage III | | |
| Renal cell carcinoma stage IV | | |
| Rhabdoid tumour of the kidney | | |

| Phimosis | Photosensitivity |
|-------------------|-----------------------------------------------|
| Acquired phimosis | Actinic elastosis |
| Phimosis | Actinic prurigo |
| | Administration site photosensitivity reaction |
| | Application site photosensitivity reaction |
| | Chronic actinic dermatitis |
| | Hartnup disease |
| | Implant site photosensitivity |
| | Infusion site photosensitivity reaction |
| | Injection site photosensitivity reaction |
| | Juvenile spring eruption |
| | Medical device site photosensitivity |
| | Photodermatosis |
| | Photokeratitis |
| | Photoonycholysis |
| | Photosensitivity reaction |
| | Polymorphic light eruption |
| | Solar dermatitis |
| | Solar urticaria |
| | Sunburn |
| | Vaccination site photosensitivity |

| Renal Related | Severe Hypersensitivity/Cutaneous AEs | Upper UTI |
|---|---|---|
| Acute kidney injury | Acute generalised exanthematous pustulosis | Bacterial pyelonephritis |
| | | Emphysematous |
| Acute phosphate nephropathy | Allergic oedema | pyelonephritis |
| Acute prerenal failure | Anaphylactic reaction | Kidney infection |
| Anuria | Anaphylactic shock | Perinephric abscess |
| Azotaemia | Anaphylactic transfusion reaction | Pyelocystitis |
| Blood creatinine increased | Anaphylactoid reaction | Pyelonephritis |
| Blood urea increased | Anaphylactoid shock | Pyelonephritis acute |
| Continuous haemodiafiltration | Angioedema | Pyelonephritis chronic |
| Dialysis | Circulatory collapse | Pyelonephritis fungal |
| Glomerular filtration rate | | |
| decreased | Circumoral oedema | Pyelonephritis mycoplasmal |
| Haemodialysis | Conjunctival oedema | Pyelonephritis viral |
| Haemofiltration | Corneal exfoliation | Pyonephrosis |
| Hypercreatininaemia | Corneal oedema | Renal abscess |
| Neonatal anuria | Cutaneous vasculitis | Renal cyst infection |
| Nephritis | Dermatitis bullous | Urosepsis |
| Nephropathy toxic | Dermatitis exfoliative | |
| Oliguria | Dermatitis exfoliative generalised | |
| Peritoneal dialysis | Drug eruption | |
| Prerenal failure | Drug hypersensitivity | |
| | Drug reaction with eosinophilia and systemic | |
| Renal failure | symptoms | |
| Renal failure acute | Epidermal necrosis | |
| Renal failure neonatal | Epiglottic oedema | |
| Renal impairment | Erythema multiforme | |
| Renal impairment neonatal | Exfoliative rash | |
| • | Eye oedema | |
| | Eye swelling | |
| | Eyelid oedema | |
| | Face oedema | |
| | First use syndrome | |
| | Fixed drug eruption | |
| | Gingival oedema | |
| | Gingival swelling | |
| | Gleich's syndrome | |
| | Hereditary angioedema | |
| | Hypersensitivity vasculitis | |
| | Idiopathic angioedema | |
| | Idiopathic urticaria | |
| | Kounis syndrome | |
| | Laryngeal dyspnoea | |
| | Laryngeal oedema | |
| | Laryngospasm | |
| | Laryngotracheal oedema | |
| | Limbal swelling | |
| | Lip exfoliation | |
| | Lip oedema | |
| | Lip swelling | |
| | Mucocutaneous ulceration | |
| | Mucosa vesicle | |
| | Mucosal erosion | |
| | Mucosal exfoliation | |
| | Mucosal necrosis | |
| | Mucosal ulceration | |
| | Nikolsky's sign | |
| | Oculomucocutaneous syndrome | |
| | Ocuromicocutaneous syndrome | |

| Renal Related | Severe Hypersensitivity/Cutaneous AEs | Upper UTI |
|---------------|---------------------------------------|-----------|
| | Oculorespiratory syndrome | |
| | Oedema mouth | |
| | Oedema mucosal | |
| | Oral mucosal blistering | |
| | Oral mucosal exfoliation | |
| | Orbital oedema | |
| | Oropharyngeal blistering | |
| | Oropharyngeal swelling | |
| | Palatal oedema | |
| | Penile exfoliation | |
| | Periorbital oedema | |
| | Pharyngeal oedema | |
| | Scleral oedema | |
| | Shock | |
| | Shock symptom | |
| | Skin exfoliation | |
| | Skin necrosis | |
| | Small bowel angioedema | |
| | Stevens-Johnson syndrome | |
| | Stridor | |
| | Swelling face | |
| | Swollen tongue | |
| | Throat tightness | |
| | Tongue exfoliation | |
| | Tongue oedema | |
| | Toxic epidermal necrolysis | |
| | Type I hypersensitivity | |
| | Urticaria | |
| | Urticaria cholinergic | |
| | Urticaria chronic | |
| | Urticaria papular | |
| | Urticarial vasculitis | |
| | Vaginal exfoliation | |

| UTI | Venous Thromboembolic events | Volume Depletion |
|---|---|---|
| Bladder candidiasis | Deep vein thrombosis | Blood pressure decreased |
| Cystitis | Deep vein thrombosis postoperative | Blood pressure orthostatic decreased |
| Cystitis bacterial | Embolism venous | Dehydration |
| Cystitis escherichia | Iliac vein occlusion | Diastolic hypotension |
| Cystitis gonococcal | Inferior vena cava syndrome | Dizziness postural |
| Cystitis haemorrhagic | Inferior vena caval occlusion | Hypotension |
| Cystitis interstitial | Jugular vein occlusion | Hypovolaemia |
| Cystitis klebsiella | Mesenteric vein occlusion | Hypovolaemic shock |
| Cystitis pseudomonal | Obstructive shock | Orthostatic hypotension |
| | Portosplenomesenteric venous | <b>.</b> 1 |
| Emphysematous cystitis | thrombosis | Orthostatic intolerance |
| | | Postural orthostatic tachycardia |
| Escherichia urinary tract infection | Post procedural pulmonary embolism | syndrome |
| Fungal cystitis | Postpartum venous thrombosis | Presyncope |
| Funguria | Pulmonary embolism | Shock |
| Genitourinary tract infection | Pulmonary infarction | Shock symptom |
| Streptococcal urinary tract | • | |
| infection | Pulmonary microemboli | Syncope |
| Ureter abscess | Pulmonary oil microembolism | Urine output decreased |
| Ureteritis | Pulmonary thrombosis | 1 |
| Uretheritis | Renal vein embolism | |

| UTI | Venous Thromboembolic events | Volume Depletion |
|---|---|---|
| Urethral abscess | Renal vein occlusion | |
| Urethral carbuncle | Subclavian vein thrombosis | |
| Urethral stricture post infection | Vascular occlusion | |
| Urinary bladder abscess | Venous thrombosis | |
| Urinary tract abscess | Venous thrombosis in pregnancy | |
| Urinary tract infection | Venous thrombosis limb | |
| Urinary tract infection bacterial | Visceral venous thrombosis | |
| Urinary tract infection | | |
| enterococcal | | |
| Urinary tract infection fungal | | |
| Urinary tract infection | | |
| pseudomonal | | |
| Urinary tract infection | | |
| staphylococcal | | |

### Appendix 1.5: Adverse Events with Potential Amputation Association

List of selected preferred terms included within the SOCs of infections and infestations, vascular disorders, nervous system disorders, and skin and subcutaneous tissue disorders

| Infections and Infestations Infected skin ulcer | Vascular<br>Disorders<br>Arteriosclerosis | Nervous System<br>Disorders<br>Paraesthesia | Skin and<br>Subcutaneous<br>Tissue Disorders<br>Diabetic ulcer | High Level Term (HLT) Skin and subcutaneous tissue ulcerations | |
|---|---|---|---|---|---|
| | | | | Penile ulceration | Medical device site erosion |
| Skin infection | Peripheral arterial occlusive disease | Hypoaesthesia | Neuropathic ulcer | Implant site ulcer | Ulcerated<br>haemangioma |
| Staphylococcal skin infection | Peripheral vascular disorder | Diabetic neuropathy | Fungating wound | Cytomegalovirus mucocutaneous ulcer | Incision site erosion |
| Gangrene | Peripheral artery stenosis | Neuropathy peripheral | Diabetic foot | Skin ulcer | Incision site ulcer |
| Osteomyelitis | Peripheral ischaemia | Areflexia | Diabetic neuropathic ulcer | Eyelid erosion | Vaccination site ulcer |
| Diabetic gangrene | Arterial stenosis | Hyporeflexia | Skin erosion | Implant site erosion | Fungating wound |
| Localised infection | Diabetic vascular disorder | Polyneuropathy | | Diabetic foot infection | Ecthyma |
| Wound abscess | Femoral artery occlusion | Autonomic neuropathy | | Application site erosion | Perineal ulceration |
| Wound infection | Thrombosis | Neuropathy peripheral | | Infusion site erosion | Tropical ulcer |
| Subcutaneous abscess | Poor peripheral circulation | Burning sensation | | Mycobacterium ulcerans infection | Injection site erosion |
| Abscess limb | Microangiopathy | Diabetic autonomic neuropathy | | Infusion site ulcer | Pyogenic sterile<br>arthritis pyoderma<br>gangrenosum and<br>acne syndrome |
| Staphylococcal osteomyelitis | Peripheral coldness | Peripheral sensory neuropathy | | Neuropathic ulcer | Scleroderma<br>associated digital<br>ulcer |
| Diabetic foot infection | Diabetic<br>microangiopathy | Peripheral<br>sensorimotor<br>neuropathy | | Skin ulcer haemorrhage | Vulval ulceration |
| Staphylococcal skin infection | Arterial occlusive disease | Sensory disturbance | | Burn infection | Mucocutaneous ulceration |
| Soft tissue infection | Arterial thrombosis | Diabetic neuropathic ulcer | | Diabetic foot | Injection site ulcer |
| Bone abscess | Peripheral artery thrombosis | | | Diabetic ulcer | Pyoderma<br>gangrenosum |
| Osteitis | Arterial occlusive disease | | | Catheter site erosion | Scrotal ulcer |
| Cellulitis | Angiopathy | | | Pyostomatitis vegetans | Application site ulcer |
| Wound <sup>a</sup> | Intermittent claudication | | | Catheter site ulcer | Genital ulceration |
| Dry gangrene | Arterial disorder | | | Medical device site ulcer | Infected skin ulcer |
| Post-operative wound infection | Impaired healing <sup>a</sup> | | | Administration site ulcer | Diabetic neuropathic ulcer |
| Post-operative wound complication a | | | | Instillation site erosion | Varicose ulceration |
| Wound dehiscence | | | | Breast ulceration | Vaginal ulceration |
| Burn infection | | | | Instillation site ulcer | Vulvovaginal ulceration |
| Extremity necrosis | | | | Administration site erosion | Auditory meatus external erosion |
| | | | | Vasculitic ulcer | Skin erosion |
| | | | | Vaccination site erosion | |

<sup>&</sup>lt;sup>a</sup> Although these PTs belong in the SOC of Injury, Poisoning and Procedural Complications or in the SOC of General Disorders and Administration Site Conditions, these terms were retained for the search strategy because of their relevance

# List of preferred terms classified as reversible infections, irreversible infections and osteomyelitis

| <b>Reversible Infections</b> | Irreversible Infections | Osteomyelitis |
|---|---|---|
| Abscess limb | Diabetic gangrene | Bone abscess |
| Burn infection | Dry gangrene | Osteitis |
| Cellulitis | Extremity necrosis | Osteomyelitis |
| Diabetic foot infection | Gangrene | Staphylococcal osteomyelitis |
| Infected skin ulcer | | |
| Localised infection | | |
| Skin infection | | |
| Soft tissue infection | | |
| Staphylococcal skin infection | | |
| Subcutaneous abscess | | |
| Wound | | |
| Wound abscess | | |
| Wound dehiscence | | |
| Wound infection | | |

50